CLINICAL TRIAL: NCT03175822
Title: Effects of Visual Art Training on Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Melody Wiseheart, Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YorkU-AD2
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Teacher
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual Arts Training (Experimental): Visual Arts Training
  Interventions: Behavioral: Visual Arts Training
- Waitlist Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Visual Arts Training — The art training program has been designed as a drawing program and focuses on basic visual art concepts (the elements [e.g., colour and line] and principles [e.g., proportion and balance] of design). Each week has a different activity and a different focus (one activity per week focusing on one element and principle of design). Each art training program will occur one hour per day, two days per week, for eight weeks. The art training program will take place at the participants' respective dementia care location in an area separate from waitlist control participants and uninvolved clients. All art programs are free for participants.
  Arms: Visual Arts Training

SUMMARY:
The purpose of the proposed study is to better understand what benefits visual art has on reducing problematic symptoms in dementia patients, including those with Alzheimer's disease.

DETAILED DESCRIPTION:
Participants:

Participants will be residents, attendees and/or members of assisted living locations and/or dementia (or related) day programs. There will be two groups: an art training group and a waitlist control group.

Data Analysis:

1. For primary measures, t-tests on pre-post difference scores comparing art training and waitlist groups.
2. For possible confounding effects, tests for confounds related to background factors (socioeconomic status, education level, gender, activity participation).

Procedure:

A randomized controlled trial design will be utilized to assess two groups of dementia patients: an art training experimental group and a structured usual-activity waitlist control group. The experimental group will participate in a visual art training program and the waitlist control group will participate in their usual structured group activities. The waitlist control group will receive the art training program once post-testing is complete. Before, during, and/or after the art programs and/or control activities, participants will be observed and complete assessments.

ELIGIBILITY:
Inclusion Criteria:

* Dementia

Exclusion Criteria:

* Inability to participate in the art training program due to physical or cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in cognition | baseline up to three weeks prior, and final assessment one to two weeks post-intervention
  Montreal Cognitive Assessment (MoCA; Nasreddine, 2005)
Change in visual working memory | baseline up to three weeks prior, and final assessment one to two weeks post-intervention
  Body Part Pointing Test (Stopford et al., 2010)
Change in auditory working memory | baseline up to three weeks prior, and final assessment one to two weeks post-intervention
  Digit Span (Weschler, 2008)

CONTACTS AND LOCATIONS:
Locations (1):
- Alzheimer's Society of York Region, Aurora, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnson KG, D'Souza AA, Wiseheart M. Art Training in Dementia: A Randomized Controlled Trial. Front Psychol. 2020 Dec 15;11:585508. doi: 10.3389/fpsyg.2020.585508. eCollection 2020. PMID 33384640